CLINICAL TRIAL: NCT05815563
Title: Validation of Peripheral Perfusion Index in Predicting Successful Supraclavicular Brachial Plexus Block for Upper Extremity Procedures in Children.
Brief Title: Validation of Peripheral Perfusion Index in Predicting Successful Supraclavicular Brachial Plexus Block in Pediatrics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed abdelghany ali, Lecturer of anesthesia, Cairo University
Other Study IDs: MD2021
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Pediatrics; Anesthesia, Local

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Few data are available for the PI as a tool for evaluation of peripheral block success in pediatric patients. Furthermore, there is currently no cut-off value defined for the accuracy of the PI in the detection of successful block.

DETAILED DESCRIPTION:
modify plan for intraoperative and postoperative analgesia. Perfusion index is an assessment of the pulsatile strength at a monitoring site; it is calculated by means of pulse oximetry by expressing the pulsatile signal as a percentage of the non pulsatile signal by a specialized probe, both of which are derived from the amount of infrared light absorbed.PI can provide useful information about the peripheral perfusion status of the patients and works as an index for sympathetic stimulation. Recent study suggested that PI could be used as an early and sensitive indicator to assess the development of sympathectomy induced by brachial plexus block in conscious adults; it is more sensitive than other parameters such as changes of skin temperature gradients or mean arterial pressure (MAP)

ELIGIBILITY:
Inclusion Criteria:

Age group: (3-14) years old. ASA class I-II

Exclusion Criteria:

* Patients with age below 3 year or older than 14 years. Parent refusal. Patients with apparent infection at site of needle insertion. Patients with any coagulation disorder. Patients with known neuropathy or brachial plexus injury. Patients with any cardiac, hepatic, renal or neurological disease

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 59 pediatric patients scheduled for elective upper extremity procedures will receive general anesthesia and trained anesthesiologist will perform ultrasound guided supraclavicular brachial plexus block on the ipsilateral side of the procedure.
Sampling Method: Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Perfusion index | Intraoperative
  The sensitivity of perfusion index in predicting success of supraclavicular brachial plexus block in pediatric patients.

SECONDARY OUTCOMES:
Temperature | Intraoperative
  The sensitivity of temperature change in predicting success of supraclavicular brachial plexus block in pediatric patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo, Egypt